CLINICAL TRIAL: NCT06691711
Title: Adult-caregiver Supported Positive Psychology Intervention to Increase Resilience (ASPIRE): Developing and Refining a Caregiver-delivered Positive Psychology Intervention to Increase the Resilience of Children Who Have Experienced Adversities - Work Package 2
Brief Title: Adult-caregiver Supported Positive Psychology Intervention to Increase Resilience: Work Package 2
Acronym: ASPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norfolk and Suffolk NHS Foundation Trust (Other)
Collaborators: University of Oxford (Other); University of Sussex (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: ASPIRE WP2
Record Dates: First submitted 2023-10-11; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2023-10

CONDITIONS: Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Waitlist controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate intervention (Experimental): Those allocated to the immediate arm will be offered the ASIRE support package over a 10 week period immediately post randomisation. The caregiver will be provided with access to all module resources and supported through the programme by a trained practitioner (their ASPIRE facilitator) who offers information, advice and encouragement during the intervention period (providing up to 8 support sessions in total).
  Interventions: Behavioral: ASPIRE support package
- Waitlist (No Intervention): Participants randomised to the waitlist arm will not be denied access to any support or treatment available as part of current service provision during the waiting period. Both young people and parents/carers will be encouraged to continue engaging with any support they already receive and can be referred/self-refer to additional services as required. After the 10-week waiting period is complete, participants randomised to this arm will be offered the ASPIRE intervention as described above.

INTERVENTIONS:
Behavioral: ASPIRE support package — The ASPIRE support package has a modular structure with core modules that all participating families are encouraged to complete initially, followed by optional modules which the family is supported to select from according to their strengths and needs. Core modules provide psychoeducation for the caregiver and optional modules contain information on the selected positive psychology topic together with instructions for suggested activities to be completed by the caregiver with their child to implement evidence-based positive psychology strategies. All resources can be accessed both electronically via an online portal or via the printed resource pack. Each caregiver is supported through the programme by a trained practitioner who offers regular support sessions (up to 8 in total) to provide information, advice and encouragement. Support sessions can take place face-to-face, by video call or over the phone according to participant preference.
  Arms: Immediate intervention

SUMMARY:
The goal of this feasibility study was to investigate a new intervention designed to help parents/carers of children aged 8-12 who have experienced adversities to build their child's resilience to mental health difficulties using a 'positive psychology' approach. The research questions concerned the acceptability, feasibility and safety of the intervention.

DETAILED DESCRIPTION:
Background: Adverse Childhood Experiences (ACEs) are traumatic or stressful events before age 18 that have been linked to poor mental health across the life course. Resilience is the ability of an individual to maintain or return to a thriving state following adversity. As resilience is not a static trait, intervening to increase the resilience of children exposed to ACEs has the potential to decrease the risk of later mental health difficulties. Positive psychology interventions (i.e. interventions that aim to increase factors that have been identified as important to individual and community flourishing) have been shown to be effective in increasing resilience. However, there was not yet a positive psychology intervention designed to meet the needs of young people exposed to ACEs and their caregivers (parents/carers).

Objectives: To investigate the acceptability, feasibility and safety of a co-produced caregiver-delivered positive psychology intervention to enhance the resilience to mental health difficulties of children who have experienced ACEs.

Methods: The project was guided by a Stakeholder Research Team (SRT) comprising both adults and young people with relevant expertise-by-experience. The study was divided into two work packages. In work package 1, the researchers completed a component analysis of existing positive psychology interventions, and a qualitative study to understand the needs and preferences of young people, parents/carers and professionals. They then conducted a series of intervention development workshops to co-produce the intervention with the SRT, informed by the findings of the component analysis and qualitative study. In work package 2, the researchers carried out a waitlist-controlled feasibility study involving 12 families with a child aged 8-12 years who had experienced ACEs. Families were randomised to receive the intervention either immediately or after a 10-week waiting period and mixed methods data collected to enable us to assess the acceptability, feasibility and safety of the intervention.

ELIGIBILITY:
Inclusion criteria:

* The child's parent or carer identifies that their child has been significantly impacted by one or more Adverse Childhood Experience (ACE).
* Child is aged 8 to 12 years.
* Child is willing and able to provide informed assent to participate.
* The child's parent or carer is willing and able provide parental consent for their child's participation.
* At least one adult caregiver (aged 18+) is willing and able to provide informed consent to participate themselves.

Exclusion criteria:

* Child is currently under the care of specialist child and adolescent mental health services (CAMHS).
* There are ongoing safeguarding concerns that might have an impact on the family's ability to participate safely (e.g. ongoing abuse or neglect).
* The child or their caregiver has a learning disability that would prevent them from accessing the intervention or completing outcome measures (reasonable adjustments will be made to allow families to participate wherever possible).

In addition, professionals involved in supporting caregivers to deliver the intervention (ASPIRE facilitators) will be invited to participate as staff participants.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Intervention feasibility / fidelity of delivery | 10 weeks
  ASPIRE intervention adherence checklist
Potential risks of the intervention | 10 weeks
  Modified Edinburgh Adverse Effects of Psychological Therapy Scale
Intervention acceptability | 10 weeks
  Qualitative acceptability of the intervention from the perspective of children, caregivers and professionals, assessed via interviews and focus groups
Intervention feasibility / fidelity of delivery | 20 weeks
  ASPIRE intervention adherence checklist
Potential risks of the intervention | 20 weeks
  Modified Edinburgh Adverse Effects of Psychological Therapy Scale
Intervention acceptability | 20 weeks
  Qualitative acceptability of the intervention from the perspective of children, caregivers and professionals, assessed via interviews and focus groups

SECONDARY OUTCOMES:
Me and My Feeling Questionnaire | Post intervention (10 weeks) & 20 week follow-up for immediate arm only
  16-item measure of mental health difficulties with emotional and behavioural difficulties subscale (child completed)
The Student Resilience Survey | Post intervention (10 weeks) & 20 week follow-up for immediate arm only
  47-item measure measuring children's perceptions of their internal and external resilience (child completed)
Students' Life Satisfaction Scale | Post intervention (10 weeks) & 20 week follow-up for immediate arm only
  7-item measure of global life satisfaction (child completed)
Strengths and Difficulties Questionnaire (parent-report version) | Post intervention (10 weeks) & 20 week follow-up for immediate arm only
  25-item measure of caregiver perception of their child's emotional and behavioural difficulties (parent/carer completed)
Me as a Parent | Post intervention (10 weeks) & 20 week follow-up for immediate arm only
  16-item measure of parental self-regulation, including their self-efficacy, personal agency, self-management and self-sufficiency as a parent (parent/carer completed)
Short Warwick Edinburgh Mental Wellbeing Scale | Post intervention (10 weeks) & 20 week follow-up for immediate arm only
  7-item measure of the parent or carer's mental wellbeing (parent/carer completed)

CONTACTS AND LOCATIONS:
Locations (1):
- Norfolk and Suffolk NHS Foundation Trust, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: No